CLINICAL TRIAL: NCT00423397
Title: A Phase I/II Pilot Study of Bioimmunotherapy With IRESSA (Gefitinib) and Pegylated Interferon Alpha-2a for Patients With Unresectable/Metastatic Squamous Cell Carcinoma of the Skin
Brief Title: Gefitinib and PEG-Interferon Alfa-2a in Treating Patients With Unresectable or Metastatic Skin Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000521454; UCSD-051205; ZENECA-IRUSIRES0488
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2008-03

CONDITIONS: Non-melanomatous Skin Cancer
Keywords: squamous cell carcinoma of the skin; recurrent skin cancer
MeSH Terms: conditions — Skin Neoplasms | interventions — peginterferon alfa-2a; Gefitinib

INTERVENTIONS:
Biological: PEG-interferon alfa-2a
Drug: gefitinib

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. PEG-interferon alfa-2a may interfere with the growth of tumor cells and slow the growth of skin cancer. Giving gefitinib together with PEG-interferon alfa-2a may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of PEG-interferon alfa-2a when given together with gefitinib and to see how well they work in treating patients with unresectable or metastatic skin cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the tolerability of gefitinib and PEG-interferon alfa-2a in patients with unresectable or metastatic squamous cell carcinoma of the skin.
* Determine the response rate in patients treated with gefitinib for 1 month.
* Determine whether the addition of weekly PEG-interferon alfa-2a to ongoing gefitinib improves response rate in these patients .
* Determine whether PEG-interferon alfa-2a exacerbates rash in patients who have been treated with gefitinib for 1 month.

OUTLINE: This is a phase I, pilot, dose de-escalation study of PEG-interferon alfa-2a followed by an open-label, phase II study.

* Phase I: Patients receive oral gefitinib alone once daily for 4 weeks. Beginning in week 5, patients also receive PEG-interferon alfa-2a subcutaneously once weekly. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of patients receive de-escalating doses of PEG-interferon alfa-2a until a tolerable dose is determined.

* Phase II: Patients receive gefitinib and PEG-interferon alfa-2a at the tolerable dose determined in phase I.

PROJECTED ACCRUAL: A total of 16 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary squamous cell carcinoma of the skin

  * Metastatic and/or unresectable locally recurrent disease
* Measurable disease
* No curative treatment option (including resection and radiotherapy) exists or is unacceptably morbid

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Bilirubin < 1.5 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV/AIDS allowed
* Patients with other cancer diagnoses (e.g., chronic lymphocytic leukemia) are eligible provided disease is controlled and does not require active treatment
* No pre-existing medical problems or laboratory abnormalities ≥ grade 3 except renal allograft patients with chronic, stable grade 3-4 renal insufficiency who are dialysis candidates

  * Nontransplant patients with any degree of renal insufficiency allowed
* No serious medical or psychiatric illness that would preclude study compliance
* No evidence of severe or uncontrolled (≥ grade 3) systemic disease (e.g., unstable or uncompensated respiratory, cardiac, or hepatic disease)

PRIOR CONCURRENT THERAPY:

* Prior solid organ transplant allowed
* Prior cytotoxic chemotherapy and radiotherapy allowed
* More than 30 days since prior experimental cancer treatment
* No prior epidermal growth factor receptor-inhibiting drugs, including gefitinib, erlotinib hydrochloride, or cetuximab
* No concurrent radiotherapy
* No concurrent cytotoxic chemotherapy or other drugs intended to control skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Tolerability
Response rate to treatment with gefitinib alone for 1 month
Response rate to treatment with gefitinib in combination with PEG-interferon alfa-2a
Toxicity
Quantification of rash after treatment with gefitinib for 1 month and after the addition of PEG-interferon alfa-2a to gefitinib

CONTACTS AND LOCATIONS:
Overall Officials: William L. Read, MD, Study Chair — University of California, San Diego
Locations (1):
- Rebecca and John Moores UCSD Cancer Center, La Jolla, California, United States